CLINICAL TRIAL: NCT03345901
Title: PROMINENT-Eye Ancillary Study: Diabetic Retinopathy Outcomes in a Randomized Trial of Pemafibrate Versus Placebo (Protocol AD)
Brief Title: PROMINENT-Eye Ancillary Study (Protocol AD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment for the substudy did not meet the goals
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DRCR.net Protocol AD
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: pemafibrate
MeSH Terms: conditions — Diabetic Retinopathy | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pemafibrate (Experimental): .2 mg pemafibrate orally BID
  Interventions: Drug: Pemafibrate
- Placebo (Placebo Comparator): Placebo pill orally BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pemafibrate — 0.2 mg orally BID - twice daily
  Arms: Pemafibrate
Drug: Placebo — orally BID - twice daily
  Arms: Placebo

SUMMARY:
Despite improved glycemic and systemic control for many patients with diabetes, over the past several decades, diabetic retinopathy (DR) develops and progresses in a large proportion of patients, and visual loss from diabetic eye complications continues to be a leading cause of blindness in the US and other developed countries worldwide. Thus, even a modest ability to prevent DR onset or to slow DR worsening might substantially reduce the number of patients at risk for diabetes-related vision loss worldwide. Widespread use of an oral agent effective at reducing worsening of DR might also decrease the numbers of patients who undergo treatment for DR and diabetic macular edema (DME) and who are consequently at risk for side effects that adversely affect visual function. Two major studies of fenofibrate, the Fenofibrate Intervention and Event Lowering in Diabetes (FIELD) and The Action to Control Cardiovascular Risk in Diabetes (ACCORD)-eye study, have demonstrated clinically important reduction in progression of retinopathy in patients with diabetes assigned to fibrate compared with placebo. However, despite the positive clinical trial results, fenofibrate has not gained wide acceptance as a preventive agent by either ophthalmologists or primary diabetes care providers. Thus, it is important to provide further evidence demonstrating whether or not selectively increasing peroxisome proliferator-activated receptor alpha (PPARα) activity reduces progression of retinopathy in patients with diabetes and non-proliferative diabetic retinopathy at baseline. Pemafibrate is a more potent and selective PPARα modulator than fenofibrate. Its efficacy is currently being evaluated in the Pemafibrate to Reduce Cardiovascular OutcoMes by Reducing Triglycerides IN patiENts With diabeTes (PROMINENT) study for prevention of cardiovascular events in patients with type 2 diabetes. Given the large study cohort with a substantial proportion likely to have DR and the multi-year duration of the PROMINENT trial, this study represents a unique opportunity to assess effects of chronic PPARα activation through pemafibrate therapy on DR outcomes.

Primary Study Objective: To assess whether treatment with pemafibrate (0.2 mg orally BID) compared with placebo reduces the hazard rate of diabetic retinopathy worsening in adults with type 2 diabetes and diabetic retinopathy without neovascularization in at least one eye who are participating in the parent PROMINENT trial.

ELIGIBILITY:
Inclusion Criteria:

* Already randomized at US or Canadian sites in the PROMINENT study
* Ability to cooperate with dilated ophthalmic examination and imaging procedures
* At least one eye meets the following study eye inclusion criteria:

  1. Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity level between 20 and 53 (minimal to severe non-proliferative diabetic retinopathy (NPDR)), inclusive, on color fundus photographs confirmed by central Reading Center grading.

Exclusion Criteria:

* Study eye exclusion criteria are:

  a. Neovascularization present. b. Current central-involved diabetic macular edema (DME based on optical coherence tomography (OCT) central subfield thickness (CST) i. Zeiss Cirrus: CST ≥ 290µm in women or ≥ 305µm in men ii. Heidelberg Spectralis: CST ≥ 305µm in women or ≥ 320µm in men c. Known major non-diabetic intraocular pathology that in the opinion of the investigator would substantially and adversely affect visual acuity or lead to ocular neovascularization during the course of the study d. Anticipated need for intravitreous anti-vascular endothelial growth factor (VEGF), intravitreous corticosteroid, or pan-retinal photocoagulation (PRP) in the next 6 months following randomization e. History of intravitreous anti-VEGF or corticosteroid treatment within the prior year for any indication.

  f. History of intraocular surgery within prior 4 months or anticipated within the next 6 months following randomization g. Any history of PRP or vitrectomy h. History of yttrium aluminum garnet (YAG) capsulotomy performed within 2 months prior to screening i. Aphakia j. Known substantial media opacities that would preclude successful imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chew, MD, Study Chair — National Eye Institute (NEI)
Locations (63):
- United States (61):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - Macula & Retina Institute, Glendale, California
  - Atlantis Eye Care, Huntington Beach, California
  - Loma Linda University Health Care, Department of Ophthalmology, Loma Linda, California
  - South Coast Retina Center, Long Beach, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retinal Consultants of Southern California Medical Group, Inc., Westlake Village, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville Health Science Cent, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Retina Macula Specialists of Miami, Miami, Florida
  - Florida Retina Institute, Orlando, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Illinois Retina Associates, S.C., Oak Park, Illinois
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - MaculaCare, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Western Carolina Clinical Research, LLC, Asheville, North Carolina
  - Kittner Eye Center, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Vitreous Center, Edmond, Oklahoma
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Retina Research Center, Austin, Texas
  - Robert E. Torti, MD, PA dba Retina Specialists, DeSoto, Texas
  - Valley Retina Institute, DeSoto, Texas
  - Retina Center of Texas, Grapevine, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Institute of Virginia, Richmond, Virginia
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin
- Canada (2):
  - UBC/VCHA Eye Care Centre, Vancouver, British Columbia
  - University Health Network - Toronto Western Hospital, Toronto

IPD SHARING:
Plan to Share IPD: Yes
Data related to the eye ancillary study will be made available after completion of the study and publication of the outcome manuscript.
Supporting Information: Study Protocol, SAP, ICF

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Participants: The study was terminated before participants were randomized to an arm. Data include all enrolled participants.
Period: Overall Study
Arm/Group | Enrolled Participants
Started | 18
Completed | 0
Not Completed | 18
Not completed — The study was terminated | 18

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 65 [54 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Diabetic Retinopathy Worsening or Diabetic Macular Edema (DME) Development (Composite Outcome)
Time Frame: 4 years
Population: The study was terminated before the participants were randomized or any study visit occurred.
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: No adverse event data were collected
Description: The study was terminated and no adverse event data were collected.
Arm/Group | Pemafibrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT03345901/Prot_SAP_000.pdf